CLINICAL TRIAL: NCT03425929
Title: Effects of a Prolonged Oxytocin Treatment on Intrusions and Amygdala Reactivity in an Analogue Trauma Model
Brief Title: Oxytocin, Trauma Disclosure and Intrusions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Rene Hurlemann, Vice Chair of the Department of Psychiatry and Chair of the Medical Psychology Division, University Hospital, Bonn
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: PROXY
Record Dates: First submitted 2018-01-28; First posted 2018-02-08 (Actual); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Healthy
Keywords: amygdala, fear, intrusion, oxytocin, trauma disclosure
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Oxytocin (6 days) (Active Comparator): Intranasal administration, 24 international units (IU) oxytocin for three days after the first trauma movie exposure and three days after the second trauma movie exposure (24 IU per day)
  Interventions: Drug: Oxytocin
- Oxytocin (3 days) (Active Comparator): Intranasal administration, 24 international units (IU) oxytocin for three days after the first trauma movie exposure (24 IU per day) and placebo nasal spray for three days after the second trauma movie exposure
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator): Placebo nasal spray for six days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — Intranasal administration, 24 international units (IU) oxytocin.
  Other Names: syntocinon
  Arms: Oxytocin (3 days); Oxytocin (6 days)
Drug: Placebo — The placebo nasal sprays contain identical ingredients except for the peptide itself.
  Arms: Placebo

SUMMARY:
Severe traumatic experiences such as falling victim to assault, torture, or rape have deleterious effects. Clinical manifestations include intrusions, avoidance behavior, and hyperarousal, which are associated, at a circuit level, with hyperfunction of the amygdala and hypofunction of prefrontal cortex (PFC) subregions. In up to 50 % of the cases, resilience is not sufficient and trauma-exposed individuals develop posttraumatic stress disorder (PTSD). Oxytocin (OXT) is a hypothalamic peptide hormone that exerts anxiolytic effects. Recent clinical trials provide preliminary evidence that post-trauma administration of OXT could be effective as a preventive intervention for PTSD in a subsample of individuals exhibiting early PTSD symptoms prior to the onset of the disorder. However, the underlying neurobiological mechanisms are unclear. Therefore, the rationale of the present project is to expose a sample of healthy participants to experimental trauma in order to explore the circuit mechanisms by which OXT influences, and interferes with, traumatic experience. Functional magnetic resonance imaging (fMRI) will be employed in order to elucidate the long-term effects of intranasal OXT on trauma-induced intrusions, amygdala and PFC responses during an emotional face matching task and resting state functional connectivity.

DETAILED DESCRIPTION:
Participants will be exposed to an experimental trauma (i.e. a highly aversive movie) at days 1 and 4 of the study. After the first experimental trauma and after the first functional magnetic resonance imaging (fMRI) measurement, the participants will receive intranasal OXT or placebo in three different groups (1. OXT for six days, 2. OXT for three days and then placebo for three days, 3. placebo for six days). The same fMRI tasks will be used after the first and second trauma exposure (i.e. one measurement before the treatment and one measurement after three days of treatment).

ELIGIBILITY:
Inclusion Criteria:

* Healthy female volunteers
* Right-handed

Exclusion Criteria:

* Current or past psychiatric disease
* Current or past physical illness
* Psychoactive medication
* Hormonal contraception
* MRI contraindication (e.g. metal in body, claustrophobia)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-03-18 (Actual); Study Completion 2017-03-18 (Actual)

PRIMARY OUTCOMES:
Total number of intrusions following the first trauma movie exposure. | Three days following the first trauma movie exposure.
  The participants will be asked to complete intrusion diaries at home in the evening of the days 1 to 3. Intrusions will be defined as involuntary recollections relating to film events that appear, apparently spontaneously, in consciousness.
Total number of intrusions following the second trauma movie exposure. | Three days following the second trauma movie exposure.
  The participants will be asked to complete intrusion diaries at home in the evening of the days 4 to 6. Intrusions will be defined as involuntary recollections relating to film events that appear, apparently spontaneously, in consciousness.
Neural responses to emotional faces in the amygdala. | Neural activations will be measured with fMRI in an emotional face matching task that lasts 20 min.
  Functional magnetic resonance imaging (fMRI) will be performed to measure blood-oxygen-level dependent signal in response to emotional face stimuli. The investigators specifically plan to investigate amygdala responses to emotional faces, because pilot data indicate that neural responses to emotional faces in these regions are associated with the total number of intrusions.
Neural responses to emotional faces in the prefrontal cortex. | Neural activations will be measured with fMRI in an emotional face matching task that lasts 20 min.
  Functional magnetic resonance imaging (fMRI) will be performed to measure blood-oxygen-level dependent signal in response to emotional face stimuli. The investigators specifically plan to investigate prefrontal cortex responses to emotional faces, because pilot data indicate that neural responses to emotional faces in these regions are associated with the total number of intrusions.
fMRI resting state data | Functional data will be acquired for 6 min.
  Participants will be instructed to lie still with open eyes during the resting state measurement and not think of anything in particular.
Trauma disclosure (time spend discussing the movie) | Six days following the first trauma movie exposure.
  The intrusion diaries will contain a question for how long participants discussed the trauma movie.

SECONDARY OUTCOMES:
Changes in pupil diameter in response to the trauma movie | 2 min baseline before the trauma movie and during 15 min of the trauma movie.
  Changes in pupil diameter will be measured.
Changes in skin conductance level in response to the trauma movie | 2 min baseline before the trauma movie and during 15 min of the trauma movie.
  Changes in skin conductance level will be measured.
Changes in respiration rate in response to the trauma movie | 2 min baseline before the trauma movie and during 15 min of the trauma movie.
  Changes in respiration rate will be measured.
Salivary oxytocin concentrations | Immediately before the trauma movie, immediately after the trauma movie and 40 min after the trauma movie.
  Saliva samples will be collected before and after the trauma movie to assess changes in oxytocin concentrations.
Salivary cortisol concentrations | Immediately before the trauma movie, immediately after the trauma movie and 40 min after the trauma movie.
  Saliva samples will be collected before and after the trauma movie to assess changes in cortisol concentrations.
Questionnaire measurement of mood (PANAS) | 10 min before and 10 min after the trauma movie.
  Positive and negative affect will be assessed via self-rating questionnaire 'The Positive and Negative Affect Schedule' using a categorical 5 point scale.

CONTACTS AND LOCATIONS:
Overall Officials: René Hurlemann, MD, PhD, Principal Investigator — University of Bonn
Locations (1):
- Department of Psychiatry, University of Bonn, Bonn, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Neuromodulation of Emotion (NEMO) research group — http://renehurlemann.squarespace.com/welcome/